CLINICAL TRIAL: NCT06736366
Title: Comparative Single-dose Bioavailability Clinical Study of Two Different Coenzyme Q10 Products
Brief Title: Study With Two Coenzyme Q10 Products
Acronym: Co10_2024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Biostile d.o.o. (Unknown); QFarm s.r.l. (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate Professor, PhD, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: Q10_2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Coenzyme Q Deficiency
Keywords: single dose bioavailability; Coenzyme Q10
MeSH Terms: conditions — Coenzyme Q10 Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 (ubiquinone) (Active Comparator): Synonyms: Maltodextrin, capsule (HPMC - hydroxypropyl methyl cellulose), coenzyme Q10 (ubiquinone); Dosage: 2 capsules, total 100 mg Co-Q10
  Interventions: Dietary Supplement: Dietary supplement - Experimental product
- BMT® coenzyme Q10 (Experimental): Maltodextrin, BMT® coenzyme Q10 [maltodextrin, coenzyme Q10 (ubiquinone), stabiliser (gum arabic), corn starch, olive oil, anti-caking agent (silicon dioxide), acidity regulators (acetic acid, citric acid)], capsule (HPMC - hydroxypropyl methyl cellulose); Dosage: 2 capsules, total 100 mg Co-Q10
  Interventions: Dietary Supplement: Dietary supplement - Active comparator

INTERVENTIONS:
Dietary Supplement: Dietary supplement - Active comparator — Single dose intervention with Standard product Coenzyme Q10 (ubiquinone); 2 capsules - 100 mg total coenzyme Q10
  Arms: BMT® coenzyme Q10
Dietary Supplement: Dietary supplement - Experimental product — Single dose intervention with Experimental product; BMT® coenzyme Q10; 2 capsules - 100 mg total coenzyme Q10
  Arms: Coenzyme Q10 (ubiquinone)

SUMMARY:
The randomized, open-label, two period crossover single-dose bioavailability study with two coenzyme Q10 products

DETAILED DESCRIPTION:
The randomized, open-label, two period crossover single-dose bioavailability study with two coenzyme Q10 products will include 35 subjects who will test two different coenzyme Q10 products. Plasma concentration of coenzyme Q10 will be measured.

ELIGIBILITY:
Inclusion Criteria:

* subject informed consent form
* aged between 50 and 65 years old
* body mass for women 70± 5 kg and for men 85± 5 kg
* non-smoking
* healthy, without cardio-vascular diseases, diabetes, neurodegenerative diseases
* absence of any prescribed medication during the study
* willing to avoid a consumption of any food supplements at least 2 weeks before and during the study

Exclusion Criteria:

* cardio-vascular diseases, diabetes, neurodegenerative diseases, gastrointestinal disorders, pregnancy, breast-feeding
* intake of any food supplements within two week of the beginning of the study
* drug or alcohol abuse

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma levels of Coenzyme Q10 | At Baseline
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.
Plasma levels of Coenzyme Q10 | Four hours after consumption
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.
Plasma levels of Coenzyme Q10 | Six hours after consumption
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.
Plasma levels of Coenzyme Q10 | Twelve hours after consumption
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.
Plasma levels of Coenzyme Q10 | Twenty-four hours after consumption
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.
Plasma levels of Coenzyme Q10 | Forthy-eight hours after consumption
  Plasma levels of Coenzyme Q10 will be measured by high-performance liquid chromatography (HPLC) with electrochemical detection and a post-analytical reducing column, using a Nanospace HPLC apparatus.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Petelin, phD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No